CLINICAL TRIAL: NCT07213349
Title: Double Blind Clinical Trial of Daridorexant (Dual Orexin Receptor Antagonist) for Alzheimer Disease Prevention
Brief Title: Daridorexant for Alzheimer Disease Prevention
Acronym: PAD-DORA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Douglas Mental Health University Institute (Other)
Collaborators: Weston Family Foundation (Other)
Responsible Party: Principal Investigator, Sylvia Villeneuve, Director of the StoP-AD Centre, Douglas Mental Health University Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DARAD2025; BH-10983 (Other Grant/Funding Number: Weston Family Foundation)
Record Dates: First submitted 2025-09-24; First posted 2025-10-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease (AD)
Keywords: Prevention; Sleep; Amyloid; Tau; Cognitive decline; Dual Orexin Receptor Antagonist (DORA); Daridorexant
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain; Cognitive Dysfunction | interventions — daridorexant

STUDY DESIGN:
Intervention Model Description: This is a single site, double blinded, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Research Staff (Research Assistants, Nurse, Coordinators)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daridorexant 50 mg (Experimental)
  Interventions: Drug: Daridorexant 50 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daridorexant 50 mg — Study drug (Daridorexant 50 mg) taken orally each night 30 minutes before bedtime, for the 1 year duration of the study
  Arms: Daridorexant 50 mg
Drug: Placebo — Study drug (Placebo) will be taken orally each night, 30 minutes before bedtime, for the 1 year duration of the study
  Arms: Placebo

SUMMARY:
This study will evaluate whether daridorexant, a DORA sleep medication, can support brain health by promoting the clearance of proteins linked to the development and progression of Alzheimer's disease. The trial is preventive and is open to participants who do not have Alzheimer's disease dementia, regardless of whether or not they experience sleep problems.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) begins decades before symptoms with the accumulation of amyloid plaques and tau tangles, and interventions that slow or prevent this process could greatly reduce its impact. Dual orexin receptor antagonists (DORAs), drugs developed for insomnia, may help clear amyloid and tau, reduce neuroinflammation, and improve cognition through mechanisms that could be both related and unrelated to sleep quality. Early animal and human studies suggest that DORAs can alter biomarkers of Alzheimer's pathology making the orexin pathway modulation a promising strategy for Alzheimer's prevention. Daridorexant, one of the two DORAs available in Canada, stands out as a well-tolerated candidate for prevention due to its safety profile.

We want to evaluate the potential of Daridorexant for prevention of AD in this single-site, double-blind, randomized (1:1), placebo-controlled trial evaluating 50 mg of daridorexant versus placebo over 12 months in 240 participants. The primary biological outcome is the change from baseline to 12 months in the plasma ratio of phosphorylated tau181 to unphosphorylated tau181 (p-tau181/np-tau181). Secondary outcomes include changes in additional plasma biomarkers, cognitive performance, sleep parameters, and safety measures.

ELIGIBILITY:
Inclusion Criteria:

* Without dementia as determined by: MoCA >21 or MMSE > 24 or Clinical Dementia Rating <1
* Minimum of 6 years of formal education
* Stable psychoactive medication for 1 month prior to screening with no intention to change dose during treatment period
* Capacity to provide written consent in English or French

Exclusion Criteria:

* Clinical diagnosis of major neurocognitive disorder
* Unstable psychiatric condition:
* Clinically significant active suicidal ideations
* Unstable medical condition in the opinion of the investigator.
* Known or suspected history of drug or alcohol dependence or abuse within one year of the screening visit
* Currently taking a DORA
* Allergy or significant adverse reaction to DORA
* Use of benzodiazepines or z-drugs > 2 times per week in the last month.
* Use of major and moderate CYP3A4 inducers and inhibitors
* Use of strong central nervous system depressants, opioids, strong analgesics, antipsychotics, sedative antidepressants.
* Active use of cholinesterase inhibitors or memantine
* Women who are breast feeding or pregnant
* Severe obstructive sleep apnea (OSA)*
* Clinically significant non-treated rapid eye movement (REM) sleep behavior disorder, restless leg syndrome or parasomnia;
* Diagnosis of narcolepsy

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in plasma p-tau217/np-tau217 ratio | baseline up to estimated 12 months
  Biological progression as measured by p-tau217/np-tau217 ratio in plasma

SECONDARY OUTCOMES:
Change in plasma p-tau181/np-tau181 ratio | baseline up to estimated 12 months
  Biological progression as measured by p-tau181/np-tau181 ratio in plasma
Change in plasma Aβ42/Aβ40 ratio | baseline up to estimated 12 months
  Biological progression as measured by Aβ42/Aβ40 ratio in plasma
Change from baseline on Preclinical Alzheimer Cognitive Composite (PACC) score | baseline up to estimated 12 months
  Cognitive progression as measured with a modified version of the Preclinical Alzheimer Cognitive Composite (PACC) score. The PACC score is created by averaging the z-scores of several neuropsychological tests to track subtle changes, where a higher PACC z-score indicates better cognition.
Change from baseline on XpressO MoCA | baseline up to estimated 12 months
  Cognitive progression as measured with the self-administered digital XpressO MoCA medical screening tool. The maximum possible score is 100 points, with higher values suggesting better cognition.

OTHER OUTCOMES:
Change in CSF Aβ42/Aβ42 | baseline up to estimated 12 months
  Change in Aβ42/Aβ40 ratio in cerebrospinal fluid in a subset of participants
Change in sleep efficiency | baseline up to estimated 12 months
  Change in sleep efficiency as measured by EEG recordings
Change in plasma GFAP | baseline up to estimated 12 months
  Change in astroglial activation and astrocytosis as measured by glial fibrillary acidic protein (GFAP) levels in plasma.
Change in p-tau181/np-tau181 after 3-months | baseline to estimated 3 months
  Biological progression as measured by p-tau181/np-tau181 ratio at 3 months, in plasma.
Change in p-tau217/np-tau217 after 3 months | baseline up to estimated 3 months
  Biological progression as measured by p-tau217/np-tau217 ratio at 3 months, in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Villeneuve, PhD, Principal Investigator — McGill University
Locations (1):
- Centre StoP-Alzheimer (Douglas Mental Health University Institute - Research Centre), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Coded individual participant data will be shared through the StoP-Alzheimer Centre open science initiatives (Repository: registeredpreventad.loris.ca and via the Canadian Open Neuroscience Platform)
URL: https://registeredpreventad.loris.ca